CLINICAL TRIAL: NCT05289245
Title: A National Registry on Clinical Manifestations, Genetics, Interventions, and Outcomes in Chinese Patients With Cystic Fibrosis (CF-CHINA)
Brief Title: A National Registry on Chinese Patients With Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XT 02
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic fibrosis (CF) is a rare autosomal recessive disease involving multiple organs, especially the lungs and digestive organs. It is most commonly seen in Caucasians. Only a few Chinese CF patients have been described in literature, taking into account the large population of China. The main objectives of this study are to accurately evaluate the prevalence of CF, the status of disease, the diagnosis and treatment, the quality of care, and the health related outcomes in China.

ELIGIBILITY:
Inclusion Criteria:

Fulfilled WHO clinical diagnostic criteria for CF; Was in a stable phase with no respiratory infections for nearly 4 weeks; Subjects (or their guardians) signed informed consent.

Exclusion Criteria:

Patients with other bronchiectasis who did not meet the inclusion criteria; Those with severe cardiac or renal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population is from across the country of China.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2032-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in spirometry (FEV1 and FVC) of lymphangioleiomyomatosis patients. | 10 years
  Spirometry will be evaluated at baseline and through study completion, an average of 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China